CLINICAL TRIAL: NCT04874584
Title: Utilizing a Culturally Tailored Nurse Coaching Intervention to Decrease Symptom Severity and Prevent Dehydration in Patients With Metastatic Cancer
Brief Title: Culturally Tailored Nurse Coaching Study for Cancer Symptom Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Oncology Nursing Society (Other)
Responsible Party: Principal Investigator, Natasha Solle, PhD, RN, assistant research professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20201491
Record Dates: First submitted 2021-04-30; First posted 2021-05-05 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Dehydration; Symptom Cluster; Quality of Life; Self Efficacy; Chemotherapy Effect
Keywords: symptom self-management; symptom severity; emotional support
MeSH Terms: conditions — Dehydration; Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CTNSM Group (Experimental): Culturally Tailored Nurse Symptom Management group (CTNSM) - participants in the CTNSM group will receive one in-person or telehealth face-to-face education session followed by a weekly telephone call and/or text message during the first 12 weeks of standard of care chemotherapy. In addition, participants can receive standard of care chemotherapy education.
  Interventions: Behavioral: CTNSM; Behavioral: Standard of Care Chemotherapy Education
- Standard of Care (control) Group (Active Comparator): Participants in the control group will only be receiving the standard of care chemotherapy education.
  Interventions: Behavioral: Standard of Care Chemotherapy Education

INTERVENTIONS:
Behavioral: CTNSM — The Culturally Tailored Nurse-delivered telephone/text message symptom-management intervention (CTNSM) intervention is an in-person or telehealth face-to-face education session followed by a weekly telephone call and/or text message conducted for the first 12 weeks of standard of care chemotherapy .
  Arms: CTNSM Group
Behavioral: Standard of Care Chemotherapy Education — Standard of Care chemotherapy education is a one-time patient education session about general treatment-related side effects patients can experience from chemotherapy and the interventions to mitigate the symptoms.

SUMMARY:
The purpose of the study is to see whether or not a telephone/ text message intervention, delivered by a registered nurse, is helpful in managing symptoms and can also prevent dehydration caused by chemotherapy treatment when given together for patients with metastatic breast, colon, lung or prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Eligible for Chemotherapy for the first time (Previous & Ongoing hormonal only treatment allowed OR Neoadjuvant & Adjuvant chemotherapy regimens with 2+ drugs allowed)
2. > 18 years old
3. Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
4. There are no life expectancy restrictions
5. Women of child-bearing potential are allowed in the study as long as they are eligible for the chemotherapy treatment.
6. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patients on immunotherapy only will be excluded
2. Previous chemotherapy
3. Under 18 years old
4. Medically Diagnosed with a Cognitive Impairment. Rationale for excluding people with cognitive impairment is that they would not be able to fully participate in the self-management care aspects of the intervention via the telephone, nor provide informed consent.
5. No access to a telephone
6. Blind or Deaf; If subject is Hearing-impaired or illiterate, then the subject may have a family member participate as a telecommunication surrogate with them in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-10-27 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Change in MDASI scores | baseline, up to 12 weeks
  MD Anderson Symptom Inventory (MDASI) is a 19 item scale with a score range from 0-10 per symptom question that measures symptom severity plus symptom interference combined to measure total symptom burden. The higher score indicates worsening of symptoms.
Incidents of dehydration | up to 12 weeks
  Incidents of unscheduled medical visits for IV hydration

SECONDARY OUTCOMES:
change in Chronic Disease Self-Efficacy Scale (CDSES) scores | baseline, up to 12 weeks
  The CDSES is a 10 item scale with a score range from 0-10 per symptom question that measures perceived self-efficacy. The higher score indicates better perceived self-efficacy.
change in Partners in Health Scale (PIHS) scores | baseline, up to 12 weeks
  The PIHS is a 12 item scale with a score range from 0-8 per question that measures symptoms self-management. The higher score indicates better symptom self-management.
Percentage of completed call or text message | up to 12 weeks
  Feasibility will be reported as a percentage of completed calls or text messages.
Change in FACT-B Scores | baseline, up to 12 weeks
  Health Related Quality of Life (HRQoL) will be measured by the Functional Assessment of Cancer Therapy -Breast (FACT-B). FACT-B has a total scoring of 0-148 with the higher scoring indicating better HRQoL.
Change in FACT-P Scores | baseline, up to 12 weeks
  Health Related Quality of Life (HRQoL) will be measured by the Functional Assessment of Cancer Therapy -Prostate (FACT-P). FACT-P has a total scoring of 0-156 with the higher scoring indicating better HRQoL.
Change in FACT-C Scores | baseline, up to 12 weeks
  Health Related Quality of Life (HRQoL) will be measured by the Functional Assessment of Cancer Therapy -Colon (FACT-C). FACT-C has a total scoring of 0-144 with the higher scoring indicating better HRQoL.
Change in FACT-LC Scores | baseline, up to 12 weeks
  Health Related Quality of Life (HRQoL) will be measured by the Functional Assessment of Cancer Therapy -Lung Cancer (FACT-LC). FACT-LC has a total scoring of 0-144 with the higher scoring indicating better HRQoL.

CONTACTS AND LOCATIONS:
Overall Officials: Natasha Solle, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami Sylvester Comprehensive Cancer Ctr., Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Nurse-Delivered Telephone Intervention to Reduce Oral Mucositis and Prevent Dehydration — https://pubmed.ncbi.nlm.nih.gov/33600392/